CLINICAL TRIAL: NCT07017322
Title: Investigating Non-invasive Cranial Electrotherapy Stimulation for Acute Anxiety in Inpatients With Eating Disorders
Brief Title: Non-invasive Cranial Electrical Stimulation for Mealtime Anxiety in Adults With Eating Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rogers Behavioral Health (Other)
Collaborators: Electromedical Products International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBH-2025-03
Record Dates: First submitted 2025-03-31; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Eating Disorders; Anxiety
Keywords: electrotherapy stimulation; Alpha-Stim AID; cranial electrotherapy stimulation; CES; meal anxiety; Non-invasive cranial electrotherapy stimulation; Inpatient weight restoration; avoidant restrictive food intake disorder; other specified feeding or eating disorder; anorexia nervosa; bulimia nervosa; purging disorder; binge eating disorder; ARFID; OSFED; procedural anxiety
MeSH Terms: conditions — Feeding and Eating Disorders; Anxiety Disorders; Avoidant Restrictive Food Intake Disorder; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder

STUDY DESIGN:
Intervention Model Description: Open-label pilot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Alpha-Stim AID Intervention Arm (Experimental): Subjects will receive treatment as usual and non-invasive cranial electrotherapy stimulation (CES) intervention using the Alpha-Stim AID device.
  Interventions: Device: Alpha-Stim AID

INTERVENTIONS:
Device: Alpha-Stim AID — Subjects will receive non-invasive cranial electrotherapy stimulation (CES) treatment in 20-minute group sessions taking place immediately prior to breakfast, lunch, and dinner. This study uses the Alpha-Stim AID® CES device which will be set to the highest amplitude that is tolerated by the participant (with a minimum of 200 microampere (µA) and a maximum of 500 µA stimulation) at 0.5 hertz for a duration of 20 minutes per session, 3 sessions per day, for 3 separate days of stimulation (180 minutes of stimulation total).

SUMMARY:
The study is to evaluate the feasibility of using a non-invasive brain stimulation device in a sample of inpatients with eating disorders (ED). The study will help researchers evaluate whether their device protocol is practical for eating disorder inpatients as a way to manage eating disorder and anxiety symptoms. A secondary aim of the study is to evaluate preliminary effectiveness of the protocol for reducing pre-meal anxiety during the treatment, and explore effects on eating disorder symptoms over the course of the inpatient admission.

DETAILED DESCRIPTION:
Evaluate the feasibility and acceptability of a protocol for using Alpha-Stim AID® (explicitly references the patented waveform and delivery method in the Alpha-Stim AID® device manufactured and marketed by Electromedical Products International, Mineral Wells, TX) to manage acute pre-meal anxiety in eating disorder inpatients indicated by recruitment and retention, dropout reasoning, nature and frequency of patient-reported side effects, level of missing patient-reported data, staff perception and patient perception. Secondary outcomes include pre-meal anxiety rated on a 0-10 visual analogue scale, eating disorder symptom severity during the three-session protocol and across the inpatient admission using the Eating Disorder-15 assessment, and clinical impairment from disordered eating using the Clinical Impairment Assessment-Eating only version, across the same timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-30 years old at the time of enrollment
2. Enrolled in Rogers Behavioral Health Eating Disorder Recovery Program Inpatient Unit at the Oconomowoc, WI clinic location
3. Have a primary diagnosis of any DSM-5 eating disorder (anorexia nervosa, bulimia nervosa, binge eating disorder, avoidant/restrictive food intake disorder, other specified feeding or eating disorder)
4. Ability to communicate effectively using written and spoken English
5. Participant is eligible for mealtime anxiety support based on:

   * ≤ 75% meal plan compliance
   * Visible anxiety/distress during program meals
   * Engagement in compensatory behaviors or self-harm before, during, or after meals, or medical staff judge patient to be at risk of same

Exclusion Criteria:

1. Metal in the body of any kind (e.g., braces, pacemakers, metal plates or screws, intracranial electrodes, implanted devices/defibrillators, prostheses)
2. Currently taking medication that reduces seizure threshold (e.g., clomipramine)
3. Cranial pathologies (e.g., holes, plates)
4. History of seizure or black-out concussion
5. Pregnancy
6. Risk of suicide/self-harm by self-strangulation with cranial electrotherapy stimulation (CES) device judged by study medical staff
7. Participant calibrates to a stimulation level below 200 microampere (μA)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who were recruited, enrolled and completed the study | From recruitment to end of study intervention at day 3.
  The percentage of eligible patients approached for recruitment, percentage of recruited patients enrolled, and percentage of enrolled patients completing the study, each as recorded by study staff.
Patient-reported dropout reason | Anytime from enrollment to the end of study intervention at day 3.
  The patient's self-reported rationale for leaving the study prematurely (e.g., unexpected discharge from inpatient eating disorder treatment, unable to tolerate stimulation, emergent suicidality, unwilling to participate in the protocol, etc.).
Patient-reported side effects | Before the first session on days 2 and 3 of the study intervention.
  Patient-reported side effects questionnaire assessing side effects experienced from the intervention day prior.
Patient perception of acceptability as assessed by the Credibility and Expectancy Questionnaire | Baseline, Days 2 and 3 of study intervention.
  The Credibility and Expectancy Questionnaire is a 6-item self-report survey used to assess patients' belief and expectation that they will benefit from a treatment. We will use two questions from the scale to assess how much the participant believes the treatment makes sense, and how strongly they feel it will help them. It is rated on a 10-point scale with anchors 1-9 (not at all (1), somewhat (5), very (9)).
  The two questions from the CEQ will be as follows:
  1. How logical does cranial electrical stimulation for pre-meal anxiety seem?
  2. How successful do you think cranial electrical stimulation will be in reducing your pre-meal anxiety?
Percent completion of study data collection | At end of patient's participation and end of admission on inpatient unit.
  Tracking and reporting completeness of all patient-reported outcome data and study data abstracted from electronic medical records.

SECONDARY OUTCOMES:
Pre-meal anxiety on a visual analogue scale on a scale from 0-10. | Prior to each meal on intervention days 1, 2 and 3.
  A patient-reported measure of pre-meal anxiety rated on a 0-10 visual analogue scale. A score of 0 is no anxiety while a score of 10 is maximum anxiety.
Eating Disorder Symptoms using the Eating Disorder-15 (ED-15) measure | From enrollment until end of study intervention on day 3.
  Patient self-reports of eating disorder symptoms using the Eating Disorder-15 (ED-15) measure. The ED-15 includes two attitudinal subscales, scored as follows: 1) Weight & Shape Concerns = mean of items 2, 4, 5, 6, 9, and 10 (add the six scores and divide by 6), 2) Eating Concerns = mean of items 1, 3, 7 and 8 (add the four scores and - divide by 4). The Overall attitudinal score is the mean of the scores on all ten items (total the ten items and divide by 10). All items are positively scored from 0-6.
The Fear of Food Measure (FOFM) | At days 1, 2 and 3 of intervention.
  The Fear of Food Measure (FOFM) is a measure of the degree to which patients report fearing eating and food itself. Scores on the FOFM can assess if patients are improving while undergoing eating disorder treatment. The FOFM is a 23 item scale positively scored 0-5 with three attitudinal scales measuring Anxiety About Eating, Food Anxiety Behaviors (i.e., avoidance), and Feared Concerns (i.e., feared outcomes of eating). Scores on all subscales will be examined, but Food Anxiety Behaviors scores are the most directly comparable across eating disorder diagnoses (e.g., Avoidant Restrictive Food Intake Disorder (ARFID) vs. anorexia and bulimia nervosa, Other Specified Feeding or Eating Disorders (OSFED)).
Eating disorder clinical impairment rated on the Clinical Impairment Assessment - Eating only (CIA) | Days 1, 2 and 3 of intervention.
  The Clinical Impairment Assessment - Eating only (CIA) is a 16-item measure of physical, cognitive, and emotional impairment from disordered eating. Items are scored on a 0-4 scale. The Eating-only version of the measure assesses impairment specifically related to restrictive or binge eating behavior, rather than impairment from other eating disorder behaviors that are not universally applicable to all eating disorders (i.e., purging, compensatory exercise). The measure is scored by summing all items for a possible score of 0-64.
Frequency of use of mealtime interventions for anxiety | Inpatient admission to discharge (average 14 days)
  Frequency of use of mealtime interventions for anxiety. This is a study-specific measure created by summing the meals during which one or more acute anxiety interventions (acute anxiolytics, one-to-one support, reduced meal plan, or tube feeding) were used across the full inpatient stay. Obtained from the electronic medical record.
Length of stay in days in the inpatient program | Inpatient admission to discharge (average 14 days).
  The outcome is time to discharge to a lower level of eating disorder care. This analysis will exclude data from any patient discharged for medical reasons, to another inpatient program, or against medical advice. Obtained from the electronic medical record.

CONTACTS AND LOCATIONS:
Locations (1):
- Rogers Behavioral Health, Oconomowoc, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No